CLINICAL TRIAL: NCT04556110
Title: Bioequivalence Study of Oral Perindopril Tert-butylamine Tablets After Meal in Healthy Subjects With a Single-dose, Randomized, Open-lable, Four-cycle, Crossover Trial Design
Brief Title: A Study on the Bioequivalence of Perindopril Tert-butylamine Tablets Taken on After Meals in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: SZYQ-BE-2018-005
Record Dates: First submitted 2020-08-25; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Healthy
Keywords: Perindopril tert-butylamine; Bioequivalence study; After meal
MeSH Terms: interventions — perindopril tert-butylamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perindopril tert-Butylamine tablets （ Produced by Haisco） (Experimental): The trial was divided into four cycles, between of each cycle with a 14-day wash-out period.In the first cycle，subjects in experimental group took the test preparation Perindopril tert-butylamine after meal, and subjects in control group took the reference preparation ACERTIL® after meal; In the second cycle subjects in experimental group took the reference preparation ACERTIL® after meal , the trial preparation perindopril tert-butylamine was taken orally after meals for the subjects in control group ; the order of taking the medicines for the subjects in the third cycle was the same as that in the first cycle, and the taking order of the subjects in the fourth cycle was the same as that in the second cycle. A single oral administration was used for the four cycles, and the dose was 4 mg.
  Interventions: Drug: Perindopril tert-Butylamine tablets （ Produced by Haisco）
- Perindopril tert-Butylamine tablets（ACERTIL®） (Active Comparator): The trial was divided into four cycles, between of each cycle with a 14-day wash-out period.In the first cycle，subjects in experimental group took the test preparation Perindopril tert-butylamine after meal, and subjects in control group took the reference preparation ACERTIL® after meal; In the second cycle subjects in experimental group took the reference preparation ACERTIL® after meal , the trial preparation perindopril tert-butylamine was taken orally after meals for the subjects in control group ; the order of taking the medicines for the subjects in the third cycle was the same as that in the first cycle, and the taking order of the subjects in the fourth cycle was the same as that in the second cycle. A single oral administration was used for the four cycles, and the dose was 4 mg.
  Interventions: Drug: Perindopril tert-Butylamine tablets（ACERTIL®）

INTERVENTIONS:
Drug: Perindopril tert-Butylamine tablets （ Produced by Haisco） — The trial was divided into four cycles, between of each cycle with a 14-day wash-out period.In the first cycle，subjects in experimental group took the test preparation Perindopril tert-butylamine after meal, and subjects in control group took the reference preparation ACERTIL® after meal; In the second cycle subjects in experimental group took the reference preparation ACERTIL® after meal , the trial preparation perindopril tert-butylamine was taken orally after meals for the subjects in control group ; the order of taking the medicines for the subjects in the third cycle was the same as that in the first cycle, and the taking order of the subjects in the fourth cycle was the same as that in the second cycle. A single oral administration was used for the four cycles, and the dose was 4 mg.
  Arms: Perindopril tert-Butylamine tablets （ Produced by Haisco）
Drug: Perindopril tert-Butylamine tablets（ACERTIL®） — The trial was divided into four cycles, between of each cycle with a 14-day wash-out period.In the first cycle，subjects in experimental group took the test preparation Perindopril tert-butylamine after meal, and subjects in control group took the reference preparation ACERTIL® after meal; In the second cycle subjects in experimental group took the reference preparation ACERTIL® after meal , the trial preparation perindopril tert-butylamine was taken orally after meals for the subjects in control group ; the order of taking the medicines for the subjects in the third cycle was the same as that in the first cycle, and the taking order of the subjects in the fourth cycle was the same as that in the second cycle. A single oral administration was used for the four cycles, and the dose was 4 mg.
  Arms: Perindopril tert-Butylamine tablets（ACERTIL®）

SUMMARY:
In order to evaluate the bioequivalence of the test preparation and reference preparation of perindopril tert-butylamine tablets after meal and their safety in Chinese adult healthy subjects.

DETAILED DESCRIPTION:
This single-center, randomized, open, single-dose, four-cycle，cross-over design bioequivalence test was conducted in subjects after meal conditions. Subjects were fasted for at least 10 hours over the night in each cycle，but can't ban their from drinking water.The next morning，after eating a high-fat and high-calorie meal for 30 minutes, according to test-reference (TR) or Reference-test (RT) sequential oral perindopril tert-butylamine tablets (4 mg, 240 mL warm water). Each period was separated with a 14-day wash-out period in after meal trials. The blood concentrations of perindopril and perindoprilat in qualified subjects were tested. Safety assessment includes vital signs examination, physical examination, laboratory safety examination, coagulation examination, electrocardiogram and adverse event reports.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers between the ages of 18 and 50 (including cut-off values), both male and female;
2. Male weight ≥50kg, female weight ≥45kg, and body mass index (BMI) 19-26kg/m2 (including cut-off values);
3. Sign the informed consent form voluntarily;
4. Be able to maintain good communication with researchers and comply with various requirements of clinical trials.

Exclusion Criteria:

1. People who is addicted to alcohol, tobacco,(drink 14 units of alcohol per week within the first month of enrollment: 1 unit = 285 ml of beer, or 25 ml of spirits, or 1 glass of wine; average daily smoking in the 3 months before screening ≥5) and/or those who cannot ban smoking and alcohol during the trial; or those who have a positive result alcohol breath trial;
2. Use any prescription drugs (such as antihypertensive drugs) within 4 weeks before screening, or use any over-the-counter drugs (vitamins, Chinese herbal tonics) within 2 weeks before screening, or take foods that affect metabolism within 2 weeks before screening, such as grapefruit or a drink containing grapefruit (acetaminophen can be used, but it must be recorded in the concomitant medication of CRF); or the subject refused to stop using foods that affect CYP1A2 during the trial, such as coffee, tea, cola, chocolate, etc.
3. Those who have used any drugs with a long half-life that may affect this study, or have participated in any drug clinical trials as subjects in the past 3 months;
4. Blood donation or blood loss ≥ 400mL within 8 weeks before the first administration;
5. People with a history of food or drug allergy, or allergies;
6. Any clinically significant physical examination, vital signs, electrocardiogram or clinical laboratory measurement abnormalities during screening;
7. Suffer from blood system, circulatory system, digestive system, urinary system, respiratory system, nervous system, immune system, endocrine system, mental abnormality, metabolic abnormality or any other chronic or serious disease history or existing disease that may affect the results of the study Those with the aforementioned systemic diseases;
8. Human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or Treponema pallidum antibody (TPPA) has a positive result;
9. Those who have a history of drug abuse or drug dependence;
10. People who have a history of fainting needles and blood, or who cannot tolerate venipuncture blood sampling and known serious bleeding tendency;
11. Patients with resting systolic blood pressure ≤90 mmHg, ≥140mmHg, or diastolic blood pressure ≤60 mmHg, ≥90mmHg, or pulse (HR) ≤50bpm, ≥100bpm;
12. Pregnant or lactating women, or female subjects whose pregnancy test results are positive; subjects (or their partners) have birth plans or sperm and egg donors during the entire trial period and within 3 months after the end of the study; trial Those who are unwilling to take one or more physical contraceptive measures during the period and within 3 months after the end of the study;
13. Patients with congenital galactosemia, glucose and galactose malabsorption syndrome, or lack of lactase;
14. Subjects who have poor compliance or who the researcher thinks are not suitable for inclusion in the group.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Maximum drug concentration (Cmax) of Perindopril | Before administration (within 2 hours) and 10 minutes to 72 hours after administration
Area under the plasma concentration versus time curve （AUC0-∞、AUC0-t）of Perindopril | Before administration (within 2 hours) and 10 minutes to 72 hours after administration

SECONDARY OUTCOMES:
Time to reach maximum plasma concentration(Tmax) of Perindopril and Perindoprilat | Before administration (within 2 hours) and 10 minutes to 72 hours after administration
Terminal elimination half-life（t1/2 ）of Perindopril and Perindoprilat | Before administration (within 2 hours) and 10 minutes to 72 hours after administration
Maximum drug concentration (Cmax) of Perindoprilat | Before administration (within 2 hours) and 10 minutes to 72 hours after administration
Area under the plasma concentration versus time curve （AUC0-∞、AUC0-t）of Perindoprilat | Before administration (within 2 hours) and 10 minutes to 72 hours after administration

OTHER OUTCOMES:
Adverse event rate | from the screening to 46 days post-dose
  Adverse events are summarized according to the system organ classification and standard name, and the system organ classification and standard name are arranged in descending order of the frequency of the tested preparation group

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of the northern theater of the Chinese people's Liberation Army, Shenyang, Liaoning, China